CLINICAL TRIAL: NCT03260998
Title: ECG Changes in Children and Adolescents With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Nagieb, principal investigator, Assiut University
Other Study IDs: ECGCCATD
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic patients type 1: electrocardiogram will be done for 60 children and adolescents with type 1 diabetes
  Interventions: Diagnostic Test: electrocardiogram
- healthy persons: electrocardiogram will be done for 60 age and sex matched non diabetic children and adolescents
  Interventions: Diagnostic Test: electrocardiogram

INTERVENTIONS:
Diagnostic Test: electrocardiogram — measurment of QT dispersion and corrected QT and other electrocardiogram changes

SUMMARY:
Diabetes Mellitus type 1 is characterized by an absolute insulin deficiency caused by T-cell-mediated autoimmune destruction of pancreatic β-cells . It is the predominant form of diabetes mellitus during childhood and adolescence. Hyperglycemia is a major cause of vascular and neuropathic complications that are seen in patients with diabetes mellitus type 1.

DETAILED DESCRIPTION:
Cardiovascular risk factors remain the most controversial chronic complication in diabetes mellitus type 1 Neuropathy in diabetes mellitus type 1 can lead to abnormalities in the response of the coronary vasculature to sympathetic stimulation, which may manifest clinically as resting tachycardia or bradycardia, exercise intolerance, orthostatic hypotension, loss of the nocturnal decline in blood pressure, or silent myocardial ischemia on cardiac testing. These abnormalities can lead to delayed presentation of cardiovascular disease. An early indicator of cardiac autonomic neuropathy is reduced heart rate variability, which can be assessed qualitatively in the clinic. Limited data suggest silent myocardial ischemia is more common in the presence of cardiac autonomic neuropathy . Cardiovascular mortality is a leading cause of death in Type 1 diabetic patients, in particular in patients with nephropathy.QT dispersion defined as the difference between maximal and minimal QT intervals from different electrocardiogram leads ( the QT interval was defined as the time between the first deflection from the isoelectric PR interval and the visual return of the T wave to the T-P segment ) ,Because these electrocardiogram abnormalities may confer an increased risk of ventricular arrhythmias and sudden cardiac death , early identification may have prognostic value .

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents with type 1 diabetes

Exclusion Criteria:

1. Cornary artery disease .
2. Heart failure , congenital heart disease ,
3. Rheumatic valve disease .
4. Primary cardiomyopathy .
5. Thyroid dysfunction .
6. Bundle branch block and atrioventricular conduction abnormalities .
7. Anti arrhythmic drugs .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 60 children and adolescents with type 1 diabetes attending Assiut university hospital and 60 sex and age matched control subjects .
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
corrected QT dispersion | one day
  difference between maximal and minimal corrected QT intervals from different ECG leads

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Atef, master, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided